CLINICAL TRIAL: NCT07277868
Title: Effect of Scapular Stabilization Exercises on Functional Outcomes in the Treatment of Subacromial Impingement Syndrome: A Controlled Clinical Study
Brief Title: Effect of Scapular Stabilization Exercises on Pain and Functional Outcomes in Subacromial Impingement Syndrome: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Karakuzu Güngör, Specialist in Physical Medicine and Rehabilitation, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: impingement-2025
Record Dates: First submitted 2025-11-27; First posted 2025-12-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Exercise Therapy; Shoulder Rehabilitation; Scapular Stabilization; Functional Outcomes
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants are allocated into two distinct groups: (1) standard physiotherapy and (2) standard physiotherapy plus scapular stabilization-mobilization-based rehabilitation.
Masking Description: The study uses single-blind masking. Only outcome assessors and statisticians are blinded to group assignments. Participants and treating physiotherapists are not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Physiotherapy (Active Comparator): Participants in this arm receive standard physiotherapy consisting of electrotherapy, range-of-motion exercises, and stretching. The program is administered three times per week for 12 weeks. No scapular-specific stabilization or mobilization exercises are included. All participants also receive a home exercise program for daily stretching and mobility exercises.
  Interventions: Other: Standard Physiotherapy
- Scapular Stabilization + Mobilization-Based Rehabilitation (Experimental): Participants receive the same standard physiotherapy as the control group, combined with a supervised scapular stabilization and mobilization-based rehabilitation program. This structured 12-week protocol (3 sessions per week) includes passive scapular mobilization (10-12 minutes per session) and a three-phase stabilization exercise progression targeting scapular mechanics, muscle activation, strength, and neuromuscular control. A daily home exercise program is also provided.
  Interventions: Other: Standard Physiotherapy

INTERVENTIONS:
Other: Standard Physiotherapy — Standard physiotherapy consisting of electrotherapy modalities, range-of-motion exercises, and stretching exercises. The program is administered three times per week for 12 weeks. The intervention does not include any scapular-specific stabilization or mobilization techniques. All participants receive a home exercise program including daily stretching and mobility exercises.
  Other Names: Conventional Physiotherapy, Routine Physiotherapy

SUMMARY:
This randomized controlled study aims to evaluate the effects of scapular stabilization exercises on pain, shoulder function, and quality of life in patients with subacromial impingement syndrome. Participants will be randomly assigned to either a scapular stabilization exercise program or a conventional shoulder rehabilitation program. Pain, functional outcome measures, and patient-reported quality of life will be assessed at baseline, 4 weeks, and 12 weeks. The study seeks to determine whether adding scapular stabilization exercises provides superior clinical benefit.

DETAILED DESCRIPTION:
Subacromial impingement syndrome (SIS) is one of the most common causes of shoulder pain and functional limitation. Scapular dyskinesis plays a key role in the development and persistence of SIS by altering scapulohumeral rhythm and increasing mechanical stress on subacromial tissues. Scapular stabilization exercises are increasingly used to restore normal scapular mechanics, improve muscular control, and reduce pain, but the clinical effectiveness of these exercises compared to conventional rehabilitation programs remains unclear.

This prospective, single-blind randomized controlled study investigates the effects of a scapular stabilization exercise program on pain, functional outcomes, and quality of life in patients diagnosed with SIS. Participants are randomly allocated to either a scapular stabilization group or a conventional shoulder rehabilitation group. Pain (VAS), functional status (QuickDASH and SPADI), range of motion, and quality-of-life measures are assessed at baseline, 4 weeks, and 12 weeks. The study aims to determine whether adding scapular stabilization exercises to standard rehabilitation leads to superior clinical improvement compared to conventional therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Clinically diagnosed subacromial impingement syndrome (SIS) based on:positive Neer test ,positive Hawkins-Kennedy test ,painful arc between 60°-120°,pain during resisted shoulder tests
* Symptoms present for at least 4 weeks.
* Ability to comply with a 12-week supervised rehabilitation program.
* Ability to provide written informed consent.

Exclusion Criteria:

* Previous shoulder surgery on the affected side.
* Presence of full-thickness rotator cuff tear confirmed by ultrasound imaging.
* Evidence of cervical radiculopathy or significant cervical spine pathology.
* Advanced glenohumeral or acromioclavicular osteoarthritis.
* History of inflammatory rheumatic diseases (e.g., rheumatoid arthritis, ankylosing spondylitis).
* Severe cardiopulmonary, neurological, or systemic conditions limiting physical activity.
* Recent shoulder fracture or dislocation (< 6 months).
* Participation in another structured shoulder rehabilitation program within the last 3 months.
* Pregnancy.
* Inability to understand or follow instructions required for the intervention or assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
1. Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) Score | Baseline, Week 6, Week 12
  QuickDASH is an 11-item validated questionnaire that measures physical function and symptoms related to upper extremity disorders. Total scores range from 0 to 100, with higher scores indicating greater disability. The primary outcome is the change in QuickDASH score from baseline to Week 12.

SECONDARY OUTCOMES:
Modified Constant-Murley Score (CMS) | Baseline, Week 6, Week 12
  The Constant-Murley Score assesses shoulder pain (15 points), daily activities (20 points), range of motion (40 points), and strength (25 points). Total score ranges from 0 to 100, with higher scores indicating better function. The secondary outcome is the improvement in CMS over time.
Visual Analog Scale (VAS) | Baseline, Week 6, Week 12
  Pain intensity at rest is measured using a 10-cm Visual Analog Scale (0 = no pain, 10 = worst pain). The outcome represents the change in resting pain levels over time.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karakuzu Güngör, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because data sharing is not planned for this study.